CLINICAL TRIAL: NCT02542813
Title: A Single Centre, Single Blind Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single Doses of Oxytocin (GR121619) Administered Via an Inhaled Route in Healthy Female Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics (PK) Study of Oxytocin (GR121619) Administered Via an Inhaled Route in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 201558
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Postpartum Hemorrhage
Keywords: Pharmacokinetics; safety; tolerability; oxytocin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IM oxytocin - IH placebo/IH oxytocin (50, 200, 400, 600) (Experimental): Subjects will receive IM oxytocin, IH placebo/IH oxytocin at doses of 50, 200, 400, 600 mcg.
  Interventions: Drug: IM oxytocin 10 IU; Drug: IH oxytocin 50 mcg; Drug: IH oxytocin 200 mcg; Drug: IH oxytocin 400 mcg; Drug: IH oxytocin 600 mcg; Drug: Placebo
- IM oxytocin - IH placebo/IH oxytocin (50) (Experimental): Subjects will receive IM oxytocin and IH placebo and/or IH oxytocin at 50 mcg.
  Interventions: Drug: IM oxytocin 10 IU; Drug: IH oxytocin 50 mcg; Drug: Placebo

INTERVENTIONS:
Drug: IM oxytocin 10 IU — IM oxytocin 10 IU is a colourless and clear sterile solution in a 1 mL ampoule containing 10 IU of oxytocin, which is administered intramuscularly
Drug: IH oxytocin 50 mcg — IH oxytocin 50 mcg is a powder blend for inhalation in a hard capsule containing 50 mcg of oxytocin, which is administered by oral inhalation.
Drug: IH oxytocin 200 mcg — IH oxytocin 200 mcg is a powder blend for inhalation in a hard capsule containing 200 mcg of oxytocin, which is administered by oral inhalation.
  Arms: IM oxytocin - IH placebo/IH oxytocin (50, 200, 400, 600)
Drug: IH oxytocin 400 mcg — IH oxytocin 400 mcg is a powder blend for inhalation in a hard capsule containing 400 mcg of oxytocin, which is administered by oral inhalation.
  Arms: IM oxytocin - IH placebo/IH oxytocin (50, 200, 400, 600)
Drug: IH oxytocin 600 mcg — IH oxytocin 600 mcg is a powder blend for inhalation in a hard capsule containing 600 mcg of oxytocin, which is administered by oral inhalation.
  Arms: IM oxytocin - IH placebo/IH oxytocin (50, 200, 400, 600)
Drug: Placebo — Placebo is a powder blend for inhalation in a hard capsule containing five inactive components, which is administered by oral inhalation.

SUMMARY:
Intramuscular (IM) oxytocin is the gold standard prophylactic therapy for post partum haemorrhage (PPH). However, in resource-poor settings within the developing world, the stability and therefore effectiveness of prophylactic IM oxytocin is diminished by a lack of appropriate refrigeration facilities and availability of trained health care professionals (HCPs) to administer IM injections. This study will be the first investigation of oxytocin in humans via the inhaled (IH) route and is designed to evaluate the safety and tolerability of inhaled oxytocin and the five non-pharmacologically active components in the placebo, and to establish the PK characteristics of up to four fixed escalating doses of inhaled oxytocin. In this single blind ascending dose-escalation study, the systemic exposure from up to four proposed escalating inhaled fixed-dose levels (50 micrograms [mcg], 200 mcg, 400 mcg and 600 mcg) will be compared with the systemic exposure following 10 international units (IU) of IM oxytocin in healthy premenopausal females.. A total of 15 subjects will be enrolled after screening sufficient number of healthy female subjects and the subjects will be assigned to one of the two treatment sequences. The total duration of this study is approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Premenopausal women on an oestrogen-containing oral contraceptive pill (OCP) for a 12 month minimum period and to continue their current OCP schedule for the duration of the clinical study and until completion of the follow-up visit.
* Physically capable of using an oral inhalation dry powder inhaler (DPI) device without physical assistance.
* FEV1.0 within normal range at screening.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body mass index (BMI) within the range 18 - 30 kilogram (kg)/square meter (m^2) (inclusive).
* Only females may participate. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: The investigator is responsible for ensuring that subjects are reminded during the study of the importance of maintaining compliance to oral contraception.
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Postmenopausal female as defined by gynaecological history.
* Chronic lung condition of any aetiology including adult asthma, chronic obstructive pulmonary disease (COPD), emphysema and interstitial lung diseases.
* Previous or current clinical history of proven pulmonary or systemic tuberculosis (TB).
* Proven or suspected respiratory tract infection / pneumonia of any aetiology within 4 weeks of screening.
* Current history of smoking and previous smokers within one year of the screening visit (if unsure about cessation of smoking status please refer to guidance below in "Relevant Habits".
* History of pulmonary embolus, pulmonary hypertension of any aetiology, and peripheral venous thromboembolism.
* Average baseline systolic blood pressure (SBP) <=100 millimeter of mercury (mmHg) at three separate readings.
* Use of an intrauterine device (IUD) within last 3 months.
* Any pregnancy within last 12 months.
* Gynaecological disorders or other diseases which can increase the risk of pelvic fibrosis are excluded, since acute uterine rupture after administration of oxytocin in postpartum women has been associated with a history of Caesarean section, possibly caused by intrauterine / pelvic scarring: a) Previous ectopic pregnancy, b) Previous pelvic, abdominal or lower spinal radiotherapy for any indication, c) Previous laparotomy for any abdominal or gynaecological indication, except no more than two previous caesarean-section(s), Previous gynaecological or urological history including endometrosis, adenomyosis, fibroids, or local bladder surgery.
* ALT and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval using Fridericia's formula (QTcF) >450 millisecond (msec) (based on triplicate ECGs).
* Prescription or non-prescription drugs not approved by the investigator, including vaginal prostaglandins within two weeks of dosing.
* History of regular alcohol consumption within 6 months of the study defined as: For United Kingdom (UK) sites: an average weekly intake of >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History or regular use of tobacco- or nicotine-containing products within one year prior to screening. Confirmatory use via a Smokerlyzer is at the discretion of the local investigator, but is advised if the subject's recent smoking history is in doubt.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation such as - Allergy to latex; allergy to any previous inhaler use.
* Positive pregnancy test at screening.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2015-12-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Up to 16 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Absolute values and changes over time of haematology from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Hematology assessments will be performed for the following parameters: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, white blood cells (WBC) (absolute), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Absolute values and changes over time of clinical chemistry from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Clinical chemistry assessments will be performed for the following parameters: blood urea nitrogen (BUN), creatinine, glucose, potassium, sodium, calcium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total and direct bilirubin, total protein, and albumin.
Absolute values and changes over time of urinalysis from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Dipstick method will be used to measure pH, glucose, protein, blood and ketones.
Absolute values and changes over time of blood pressure from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Three readings of blood pressure will be taken at screening (single readings at all other time-points).
Absolute values and changes over time of pulse rate from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Three readings of pulse rate will be taken at screening (single readings at all other time-points).
Absolute values and changes over time of heart rate from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Absolute values and changes over time of heart rate from pre-dose values as a measure of safety and tolerability.
Absolute values and changes over time of 12-lead electrocardiogram (ECG) parameters (PR, QRS, QT, corrected QT [QTc] intervals) from pre-dose values as a measure of safety and tolerability | Up to 20 weeks
  Triplicate 12-lead ECGs will be obtained screening and predose (predose IM oxytocin), and single 12-lead ECGs at all other time-points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Number of subjects with adverse respiratory events as monitored by spirometry including forced expiratory volume in 1 second (FEV1.0) and pulse oximetry as a measure of specific respiratory safety | Up to 16 weeks
  FEV1 is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. Pulse oximetry is a procedure used to measure the oxygen level (or oxygen saturation) in the blood.
Plasma concentration profile for IH oxytocin | Day 1, 2, and 3 of dosing session 1, and Day 1 of dosing session 2, 3, and 4
  Blood samples will be withdrawn from subjects at pre dose, 3 minutes (mins), 5 mins, 10 mins, 20 mins, 0.5h, 0.75h, 1 hour (h), 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 8 h, and 24 h (24 h post dose assessments only applicable to Dosing Session 1, Group 1 and the first 3 subjects at each new dose level [Dosing Sessions 2 -4]).
Plasma concentration profile for 10 IU IM oxytocin | Day 1, 2, and 3 of dosing session 1, and Day 1 of dosing session 2, 3, and 4
  Blood samples will be withdrawn from subjects at pre dose, 3 mins, 5 mins, 10 mins, 20 mins, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, and 8 h.
Composite PK parameters for IH oxytocin: maximum plasma concentration (Cmax), last quantifiable concentration (Clast), time to Cmax (tmax), area under the plasma concentration-time curve (AUC) and terminal phase half-life (t1/2) | Day 1, 2, and 3 of dosing session 1, and Day 1 of dosing session 2, 3, and 4
  Blood samples will be withdrawn from subjects at pre dose, 3 mins, 5 mins, 10 mins, 20 mins, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 8 h, and 24 h (24 h post dose assessments only applicable to Dosing Session 1, Group 1 and the first 3 subjects at each new dose level [Dosing Sessions 2 -4]).
Composite PK parameters for 10 IU IM oxytocin: Cmax, Clast, tmax, AUC and t1/2 | Day 1, 2, and 3 of dosing session 1, and Day 1 of dosing session 2, 3, and 4
  Blood samples will be withdrawn from subjects at pre dose, 3 mins, 5 mins, 10 mins, 20 mins, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, and 8 h.

SECONDARY OUTCOMES:
Composite of PK parameters: Cmax and AUC will be compared as data permit | Day 1, 2, and 3 of dosing session 1, and Day 1 of dosing session 2, 3, and 4
  For IM oxytocin: Blood samples will be withdrawn from subjects at pre dose, 3 mins, 5 mins, 10 mins, 20 mins, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, and 8 h.For IH oxytocin: Blood samples will be withdrawn from subjects at pre dose, 3 mins, 5 mins, 10 mins, 20 mins, 0.5 h, 0.75 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 8 h, and 24 h (24 h post dose assessments only applicable to Dosing Session 1, Group 1 and the first 3 subjects at each new dose level [Dosing Sessions 2 -4]).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Fernando D, Siederer S, Singh S, Schneider I, Gupta A, Powell M, Richards D, McIntosh MP, Lambert P, Fowles S. Safety, Tolerability and Pharmacokinetics of Single Doses of Oxytocin Administered via an Inhaled Route in Healthy Females: Randomized, Single-blind, Phase 1 Study. EBioMedicine. 2017 Aug;22:249-255. doi: 10.1016/j.ebiom.2017.07.020. Epub 2017 Jul 22. PMID 28781129
- See also: Results for study 201558 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201558?search=study&b'search_terms=201558'#rs
- Available data/document: Statistical Analysis Plan: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201558 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register